CLINICAL TRIAL: NCT01668849
Title: Preliminary Clinical Trial Investigating the Ability of Plant Exosomes to Abrogate Oral Mucositis Induced by Combined Chemotherapy and Radiation in Head and Neck Cancer Patients
Brief Title: Edible Plant Exosome Ability to Prevent Oral Mucositis Associated With Chemoradiation Treatment of Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Rebecca Redman, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12.0220
Record Dates: First submitted 2012-08-06; First posted 2012-08-20 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Head and Neck Cancer; Oral Mucositis
Keywords: Plant exosomes; Grape exosomes; Grape extract; Oral mucositis; Head and Neck Cancer; Immune response
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis | interventions — whole grape extract; oxycodone-acetaminophen; Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Grape extract (Experimental): Grape extract self-administered daily by mouth for 35 days during chemoradiation therapy.
  Interventions: Dietary Supplement: Grape extract
- 2 - Lortab, Fentanyl patch, mouthwash (Active Comparator): Standard oral mucositis therapy such as pain medication and anti-fungal mouth washes will be prescribed according to product labels.
  Interventions: Drug: Lortab, Fentanyl patch, mouthwash

INTERVENTIONS:
Dietary Supplement: Grape extract — Grape extract self-administered by mouth daily for 35 days
  Arms: 1 - Grape extract
Drug: Lortab, Fentanyl patch, mouthwash — Lortab 5-10 mg Fentanyl patch 25 mcgs Mary's Magic Mouthwash
  Other Names: Lortab 5-10 mg; Fentanyl patch 25 mcgs; Mary's Magic Mouthwash
  Arms: 2 - Lortab, Fentanyl patch, mouthwash

SUMMARY:
This study will evaluate the ability of grape exosomes, given to the subject as grape powder, as an important anti-inflammatory agent to reduce the incidence of oral mucositis during radiation and chemotherapy treatment for head and neck tumors.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the ability of plant (grape) exosomes to prevent oral mucositis associated with chemoradiation treatment of head and neck cancer. Also, to be evaluated is the effect of grape exosomes on the production of cytokines and immune responses to tumor exosomal antigens, metabolic and molecular markers in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have definitive diagnosis of head and neck cancer.
* Concurrent chemoradiation treatment of the primary tumor must be an option for the newly diagnosed cancer.
* Patients must be informed of the investigational nature of this study and sign and give written informed consent in accordance with institutional and federal guidelines.
* Absence of life limiting medical conditions
* Ability to understand and willingness to sign a written informed consent document.
* ECOG performance status 0, 1, or 2 (Karnofsky > 60%).
* Patients must have adequate bone marrow function. ANC > 1000/microL and Platelet count >100,000/microL
* Age >20 years

Exclusion Criteria:

* Known familial head and neck cancer syndrome
* Pregnancy
* Known HIV
* Patients receiving immunosuppressive drugs
* Inflammatory bowel disease
* Active second malignancy in the last 5 years
* Patients receiving any other investigational agent(s)
* Patients who have received any prior chemotherapy or radiation therapy to the primary head and neck cancer

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08-02 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Pain caused by oral mucositis | Total followup of six months
  Extent of pain from oral mucositis will be evaluated weekly during treatment (6 to 7 weeks) and for six months following the completion of treatment which will last approximately 30 days.

SECONDARY OUTCOMES:
Level of immune biomarkers in blood | Within three days of the completion of radiation therapy which will last approximately 30 days.
  Levels of immune biomarkers (cytokines, T cells NK Cells CD11cIL12)in the blood at the time of completion of radiation therapy will be compared to baseline levels.
Level of immune biomarkers in mucosal tissue | Within three days of the completion of radiation therapy which will last approximately thirty days.
  Levels of immune biomarkers (CD3, CD8, CD11b, F4/80, BRDU)in scrapings of mucosal tissue at the time of completion of radiation therapy will be compared to baseline levels.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Redman, MD, Principal Investigator — James Graham Brown Cancer Center, University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Wu K, Xing F, Wu SY, Watabe K. Extracellular vesicles as emerging targets in cancer: Recent development from bench to bedside. Biochim Biophys Acta Rev Cancer. 2017 Dec;1868(2):538-563. doi: 10.1016/j.bbcan.2017.10.001. Epub 2017 Oct 18. PMID 29054476
- See also: James Graham Brown Cancer Center, Louisville, Kentucky — http://www.browncancercenter.org